CLINICAL TRIAL: NCT00752063
Title: A Phase IIa Trial of Sorafenib With Capecitabine and Oxaliplatin in Patients With Locally Advanced or Metastatic Hepatocellular Carcinoma
Brief Title: Sorafenib With Capecitabine and Oxaliplatin for Advanced or Metastatic Hepatocellular Carcinoma
Acronym: SECOX
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Professor Ronnie Poon, The University of Hong Kong,
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HKU-SRG-P001
Record Dates: First submitted 2008-09-01; First posted 2008-09-15 (Estimated); Last update posted 2008-09-15 (Estimated); Status verified 2008-09

CONDITIONS: Advanced Hepatocellular Carcinoma; Metastatic Hepatocellular Carcinoma
Keywords: Sorafenib; Capecitabine; Oxaliplatin; Advanced Hepatocellular Carcinoma; Metastatic Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib; Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): All subjects will receive Sorafenib with Capecitabine and Oxaliplatin
  Interventions: Drug: Sorafenib with Capecitabine and Oxaliplatin

INTERVENTIONS:
Drug: Sorafenib with Capecitabine and Oxaliplatin — Regimen 1: Oxaliplatin 85 mg/m2 (50 mg per vial) administered intravenously on day 1 of each cycle Regimen 2: Capecitabine 1700 mg/m2 p.o. (850 mg/m2 BD) day 1 to 7 Regimen 3: Sorafenib 400 mg (200 mg/tablet) orally BD day 1 to 14

SUMMARY:
HCC is an aggressive, largely chemo-resistant cancer with a poor prognosis, currently there is no effective systemic chemotherapy for HCC. Epidermal growth factor receptor (EGFR) and vascular endothelial growth factor (VEGF) are both overexpressed in HCC and thought to contribute to tumor development. Oxaliplatin in combination with other chemotherapies or biologic agents have been shown to be an effective and safe treatment in advanced HCC patients.

Sorafenib, an oral multi-kinase inhibitor, blocks tumor cell proliferation by targeting multiple growth factor pathways and also exerts an anti-angiogenic effect. Clinically, single agent Sorafenib has been shown to have some efficacy in patients with advanced HCC and the primary result of prolonged overall survival seems to have been achieved in the phase III trial.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is the most common primary liver malignancy, with an annual incidence of over 500,000 new patients and more than half of the new cases occur in China. The most common etiological causes of HCC are hepatitis B and hepatitis C viral infections.

HCC is a cancer of high particular relevance in Hong Kong because of the high prevalence (10%) of hepatitis B virus infection in the population. It is the second most common cancer causing death in Hong Kong. Surgical resection and liver transplantation are regarded as the main curative treatments for HCC. Nevertheless, the majority of patients have unresectable HCCs because of advanced tumor stage and poor liver function. Besides, transplantation is indicated only for early small HCCs, and its application is limited by the shortage of liver graft, which is a particularly severe problem in Hong Kong.

HCC is an aggressive, largely chemo-resistant cancer with a poor prognosis, currently there is no effective systemic chemotherapy for HCC. Epidermal growth factor receptor (EGFR) and vascular endothelial growth factor (VEGF) are both overexpressed in HCC and thought to contribute to tumor development. Oxaliplatin in combination with other chemotherapies or biologic agents have been shown to be an effective and safe treatment in advanced HCC patients. Sorafenib, an oral multi-kinase inhibitor, blocks tumor cell proliferation by targeting multiple growth factor pathways and also exerts an anti-angiogenic effect.

Sorafenib has been approved by FDA for use in renal cell carcinoma based on prolonged survival in phase III trials. Single agent Sorafenib has been shown to have some efficacy in patients with advanced HCC and the primary result of prolonged overall survival have been achieved in a recent randomized phase III trial. However, most patients would only have disease stabilization as the phase II trial only showed a tumor response rate of only 8% (PR & MR). Combination with chemotherapy may improve the tumor response rate.

ELIGIBILITY:
Inclusion Criteria:

* Patients with locally advanced or metastatic HCC not suitable surgical or locoregional therapies
* Age more than 18 years
* Performance status 0 or 1
* Life expectancy of 3 months
* Prior radiotherapy more than 3 weeks prior to study entry
* No prior systemic therapy
* Hb more than 8.5 g/dl
* ANC more than 1,500/mm3
* PLT more than 75 x 109/L
* PT-INR/PTT less than 1.5 x upper limit of normal
* Total bilirubin of less than 1.5 x upper limit of normal
* Serum creatinine less than 1.5 x upper limit of normal
* Serum AST and ALT less than 2.5 x upper limit of normal

Exclusion Criteria:

* History of cardiac disease
* Symptomatic metastatic brain or meningeal tumors
* Main portal vein tumor thrombosis
* Ascites uncontrolled by medication
* Variceal or gastrointestinal bleeding within three months prior to start of treatment
* Seizure disorder requiring medication
* Patients undergoing renal dialysis
* Previous or concurrent cancer that is distinct in primary site
* Prior use of any systemic anti-cancer treatment
* Prior use of Raf-kinase inhibitors (RKI), VEGF inhibitors, MEK inhibitors or Farnesyl transferase inhibitors
* Patients on any local ablative treatment or TACE within 6 weeks
* Radiotherapy during study or within 3 weeks
* Major surgery within 4 weeks
* Concomitant treatment of rifampin or St John's Wort
* Pregnant or breast-feeding patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2007-09; Primary Completion 2008-12 (Estimated); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 4 cycles

SECONDARY OUTCOMES:
Tumor response rate, overall survival and safety of the regimen in HCC patients | 8 cycles

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Mary Hospital, Hong Kong, China